CLINICAL TRIAL: NCT06040086
Title: A Phase III, Multicentre, Randomised, Double-blind, Chronic-dosing, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Tozorakimab in Participants With Symptomatic Chronic Obstructive Pulmonary Disease (COPD) With a History of COPD Exacerbations (MIRANDA)
Brief Title: Efficacy and Safety of Tozorakimab in Symptomatic Chronic Obstructive Pulmonary Disease With a History of Exacerbations
Acronym: MIRANDA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9180C00012; 2023-505543-39-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-08-25; First posted 2023-09-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD; tozorakimab; MEDI3506; exacerbations; ICS; LABA/LAMA; Biologic; Biologic Treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tozorakimab (Experimental): Dosing subcutaneously tozorakimab
  Interventions: Drug: Tozorakimab
- Placebo (Placebo Comparator): Dosing subcutaneously with equivalent volume to tozorakimab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo administered subcutaneously, equivalent volume to tozorakimab throughout the study.
  Arms: Placebo
Drug: Tozorakimab — Administered subcutaneously tozorakimab and placebo throughout the study.
  Arms: Tozorakimab

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy and safety of tozorakimab administered subcutaneously (SC) in adult participants with symptomatic COPD with a history of ≥ 2 moderate or ≥ 1 severe exacerbations of COPD in the 12 months prior to enrolment. Participants should be receiving optimised treatment with inhaled maintenance therapy (ICS/LABA/LAMA triple therapy, or dual therapy if triple is not considered appropriate) throughout at least the last 3 months prior to enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 40 years of age and capable of giving signed informed consent.
2. Documented diagnosis of COPD for at least one year prior to enrolment.
3. Post BD FEV1/FVC < 0.70 and post-BD FEV1 >20% of predicted normal value
4. Documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbations within 12 months prior to enrolment.
5. Documented optimised inhaled dual or triple therapy for at least 3 months prior to enrolment.
6. Smoking history of ≥ 10 pack-years.
7. CAT total score ≥ 10, with each of the phlegm (sputum) and cough items with a score ≥ 2

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD.
2. Radiological findings suggestive of a respiratory disease other than COPD that is significantly contributing to the participant's respiratory symptoms. Radiological findings of pulmonary nodules suspicious for lung cancer, as per applicable guidances, without appropriate follow up prior to randomisation. Radiological findings suggestive of acute infection.
3. Current diagnosis of asthma, prior history of asthma, or asthma-COPD overlap. Childhood history of asthma is allowed and defined as asthma diagnosed and resolved before the age of 18
4. Any unstable disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric disorder, major physical and/or cognitive impairment that could affect safety, study findings or participants ability to complete the study.
5. COPD exacerbation, within 2 weeks prior to randomization, that was treated with systemic corticosteroids and/or antibiotics, and/or led to hospitalization.
6. Active significant infection within the 4 weeks prior to randomization, pneumonia within 6 weeks prior to randomization, or medical condition that predisposes the participant to infection.
7. Suspicion of, or confirmed, ongoing SARS-CoV-2 infection.
8. Significant COVID-19 illness within the 6 months prior to enrolment.
9. Unstable cardiovascular disorder.
10. Diagnosis of cor pulmonale, pulmonary arterial hypertension and/or right ventricular failure.
11. History of active severe inflammatory bowel disease or colitis within one year prior to enrolment, or unexplained diarrhoea within the 4 weeks prior to randomisation.
12. History of known immunodeficiency disorder, including a positive test for HIV-1 or HIV 2.
13. History of positive test or treatment for hepatitis B or hepatitis C (except for cured hepatitis C)
14. Evidence of active liver disease, including jaundice during screening.
15. Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than one year prior to enrolment. Suspected malignancy or undefined neoplasms.
16. Participants who have evidence of active TB.
17. History of partial or total lung resection.
18. Scheduled major surgical procedure during the course of the study.
19. Participants that have previously received tozorakimab.
20. Any clinically significant abnormal findings in physical examination, vital signs, ECG, or laboratory testing during the screening period, which in the opinion of the investigator may put the participant at risk because of their participation in the study, or may influence the results of the study, or the participant's ability to complete the entire duration of the study.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1454 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate to severe COPD exacerbations in participants who are former smokers. | Over 52 weeks
  The primary endpoint will be assessed in the primary population (former smokers with symptomatic COPD and a history of exacerbations, on optimised treatment with maintenance inhaled therapy [triple therapy, or dual therapy if triple is not considered appropriate]).

SECONDARY OUTCOMES:
Annualized rate of moderate to severe COPD exacerbations in former or current smokers. | Over 52 weeks
  The annualized rate will be assessed in the overall population of participants including current and former smokers with symptomatic COPD and history of exacerbations, on optimised treatment with maintenance inhaled therapy.
Change from baseline in SGRQ total score from in former smokers | Over 52 weeks
  Difference in mean change from baseline in SGRQ total score in former smokers.
Change from baseline in SGRQ total score from in the overall population of current and former smokers. | Over 52 weeks
  Difference in mean change from baseline in SGRQ total score in the overall population of current and former smokers.
Annualized rate of severe COPD exacerbations in former smokers | Variable duration period up to study completion, approximately 3 years
  The rate ratio of severe COPD exacerbations will be assessed in former smokers.
Annualized rate of severe COPD exacerbations in former or current smokers | Variable duration period up to study completion, approximately 3 years
  The rate ratio of severe COPD exacerbations will be assessed in the overall population of current and former smokers.
Change from baseline in E-RS:COPD total score in former smokers | Over 52 weeks
  Difference in mean change in E-RS:COPD total score from baseline in former smokers.
Change from baseline in E-RS:COPD total score in former or current smokers | Over 52 weeks
  Difference in mean change in E-RS:COPD total score from baseline in the overall population of current and former smokers.
Change from baseline in pre-bronchodilator, pre dose trough FEV1 (mL) in former smokers | Over 52 weeks
  Change from baseline in pre-bronchodilator, pre dose trough FEV1 (mL) in former smokers.
Change from baseline in pre-bronchodilator, pre dose trough FEV1 (mL) in former or current smokers | Over 52 weeks
  Change from baseline in pre-bronchodilator, pre dose trough FEV1 (mL) in the overall population of current and former smokers.
Change from baseline in post-bronchodilator FEV1 (mL) in former smokers | Week 52
  Change from baseline in post-bronchodilator FEV1 (mL) in former smokers.
Change from baseline in post-bronchodilator FEV1 (mL) in former smokers or current smokers | Week 52
  Change from baseline in post-bronchodilator FEV1 (mL) in former smokers or current smokers.
Annualised rate of COPD exacerbations requiring hospitalisations and/or Emergency Room (ER)/Emergency Department (ED) visits in former smokers | Variable duration period up to study completion, approximately 3 years
  The rate ratio of COPD exacerbations requiring hospitalisations and/or Emergency Room (ER)/Emergency Department (ED) visits in former smokers.
Annualised rate of COPD exacerbations requiring hospitalisations and/or Emergency Room (ER)/Emergency Department (ED) visits in former or current smokers | Variable duration period up to study completion, approximately 3 years
  The rate ratio of COPD exacerbations requiring hospitalisations and/or Emergency Room (ER)/Emergency Department (ED) visits in former or current smokers.
Change from baseline in pre-BD, pre-dose trough FEV1 (mL) | 52 weeks
  Change from baseline in pre-BD, pre-dose trough FEV1 (mL).
Change from baseline in post-BD FEV1 (mL) | Over 52 weeks
  Change from baseline in post-BD FEV1 (mL).
Time to first moderate to severe COPD exacerbation | Over 52 weeks
  Time to first moderate to severe COPD exacerbation compared with placebo.
Time to first severe COPD exacerbation | Variable duration period up to study completion, approximately 3 years
  Time to first severe COPD exacerbation compared with placebo.
Change from baseline in CAT total score | Week 52
  Change from baseline in CAT total score compared with placebo.
Proportion of participants achieving MCID in CAT score | Week 52
  Proportion of participants achieving MCID in CAT score (percentage of participants with a decrease in CAT total score of ≥ 2 points from baseline).
Proportion of participants achieving MCID in SGRQ total score | Week 52
  Proportion of participants achieving MCID in SGRQ score (percentage of participants with a decrease in SGRQ total score of ≥ 4 points from baseline).
Proportion of participants achieving MCID in E-RS:COPD total score | Week 52
  Proportion of participants achieving MCID in E-RS:COPD total score (percentage of participants with a decrease in E-RS:COPD total score of ≥ 2 points from baseline).
Annualized rate of healthcare resource utilization | Variable duration period up to study completion, approximately 3 years
  Annualized rate of healthcare resource utilization.
Change from baseline in rescue medication | Over 52 weeks
  Change from baseline (difference in mean number of puffs/day) in rescue medication use.
Trough serum concentrations of tozorakimab | Over 52 weeks
  Pharmacokinetics: concentrations of tozorakimab in trough serum.
Presence of anti-drug antibodies | Over 52 weeks
  Immunogenicity: presence of tozorakimab anti-drug antibodies in blood serum.
Time to death | Variable duration period up to study completion, approximately 3 years
  Time to death (all-cause mortality)

CONTACTS AND LOCATIONS:
Locations (326):
- United States (54):
  - Research Site, Birmingham, Alabama
  - Research Site, Decatur, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Yuma, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Westminster, California
  - Research Site, Aurora, Colorado
  - Research Site, Boulder, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boynton Beach, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lithonia, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Andover, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Towson, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Hannibal, Missouri
  - Research Site, Papillion, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Toms River, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Lima, Ohio
  - Research Site, Grants Pass, Oregon
  - Research Site, Gaffney, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Elizabethton, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Roy, Utah
  - Research Site, Kenosha, Wisconsin
- Argentina (11):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Belgium (8):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Mechelen
  - Research Site, Namur
  - Research Site, Roeselare
- Brazil (11):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, São Bernardo do Campo
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Valinhos
- Bulgaria (7):
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Panagyurishte
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Veliko Tanovo
  - Research Site, Yambol
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Winchester, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
- Chile (5):
  - Research Site, Chile
  - Research Site, Concepción
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Viña del Mar
- China (30):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Liaocheng
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Pingxiang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Taizhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Zigong
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Roskilde
  - Research Site, Vejle
- France (11):
  - Research Site, Aix-en-Provence
  - Research Site, Brest
  - Research Site, Colmar
  - Research Site, Epagny Metz-Tessy
  - Research Site, La Tronche
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Villefranche-sur-Saône
- Germany (18):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Moers
  - Research Site, München
  - Research Site, München-Pasing
  - Research Site, Nuremberg
  - Research Site, Peine
  - Research Site, Solingen
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- Hungary (10):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Edelény
  - Research Site, Encs
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Mosonmagyaróvár
  - Research Site, Pécs
  - Research Site, Százhalombatta
  - Research Site, Szolnok
- India (11):
  - Research Site, Ajmer
  - Research Site, Calicut
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Dwārka
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Nagpur
  - Research Site, Vijayawada
  - Research Site, Visakhapatnam
- Ireland (4):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Galway
  - Research Site, Moneymore
- Italy (8):
  - Research Site, Cona
  - Research Site, Foggia
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Roma
- Japan (50):
  - Research Site, Aomori
  - Research Site, Asahikawa-shi
  - Research Site, Chikushino-shi
  - Research Site, Chūōku
  - Research Site, Fujieda-shi
  - Research Site, Fukuoka
  - Research Site, Ginowan-shi
  - Research Site, Habikino-shi
  - Research Site, Hakodate-shi
  - Research Site, Hamamatsu
  - Research Site, Iizuka-shi
  - Research Site, Itabashi-ku
  - Research Site, Izumi-shi
  - Research Site, Kagoshima
  - Research Site, Kasuga-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawachinagano-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kiyose-shi
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Kusatsu-shi
  - Research Site, Kyoto
  - Research Site, Matsusaka-shi
  - Research Site, Minoh
  - Research Site, Minokamo Shi
  - Research Site, Mizunami-shi
  - Research Site, Morioka
  - Research Site, Nagoya
  - Research Site, Nankoku-shi
  - Research Site, Ogaki-shi
  - Research Site, Okinawa-shi
  - Research Site, Omuta-shi
  - Research Site, Osaka
  - Research Site, Sagamihara-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shizuoka
  - Research Site, Tachikawa-shi
  - Research Site, Toon-shi
  - Research Site, Toride-shi
  - Research Site, Toshima-ku
  - Research Site, Toyonaka-shi
  - Research Site, Ube
  - Research Site, Ueda-shi
  - Research Site, Urasoe-shi
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Malaysia (6):
  - Research Site, Alor Star
  - Research Site, Kajang
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Seremban
- Research Site, Mexico City, Mexico
- Netherlands (7):
  - Research Site, 's-Hertogenbosch
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Heerlen
  - Research Site, Roermond
  - Research Site, Rotterdam
  - Research Site, Zutphen
- Peru (3):
  - Research Site, Lima
  - Research Site, Piura
  - Research Site, Santa Beatriz
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Pruszków
  - Research Site, Płock
  - Research Site, Rzeszów
- South Korea (6):
  - Research Site, Anyang-si
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (8):
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Cáceres
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Santander
  - Research Site, Zaragoza
- Thailand (5):
  - Research Site, Hat Yai
  - Research Site, Khlong Luang
  - Research Site, Muang
  - Research Site, Mueang
  - Research Site, Nakhon Ratchasima
- Turkey (Türkiye) (3):
  - Research Site, Adana
  - Research Site, Istanbul
  - Research Site, Mersin
- Ukraine (8):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Tarasove Village
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (10):
  - Research Site, Bradford
  - Research Site, Cottingham
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Macclesfield
  - Research Site, Newcastle upon Tyne
  - Research Site, Portsmouth
  - Research Site, Wakefield
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at :
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/